CLINICAL TRIAL: NCT00881335
Title: Implemental Flutter Mucus Clearance Devices on Geriatric Lung Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Zhang Xiangyu, MD, director, professor, FCCM, FCCP., Tongji University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SHDC12007211-O
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Pulmonary Disease
Keywords: geriatric; pulmonary disease; flutter; sputum; physical therapy techniques
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention)
- intervention (Experimental): Intervention group were given flutter valve mucus clearance devices to do pulmonary function exercise
  Interventions: Device: flutter mucus clearance device

INTERVENTIONS:
Device: flutter mucus clearance device — five minutes every sessions, three sessions per day
  Arms: intervention

SUMMARY:
The purpose of this study is to evaluate the clinical outcome and safety of flutter mucus clearance devices in elders of gerocomium.

DETAILED DESCRIPTION:
Respiratory diseases are still increasing in the elderly population. The fluttering mucus clearance technique is expected to be a physical assisting therapy enhancing airway secretion clearance but needs more clinical randomized, controlled trial evidence.

ELIGIBILITY:
Inclusion Criteria:

* available to perform the device, the elders in geracomium
* male and female
* aging 85 years or more

Exclusion Criteria:

* not available to perform the procedure
* untreated pneumothorax
* diffusion interstitial lung disease
* acute coronary syndrome
* third stage hypertension
* advanced cancer
* severe heart, liver, renal, blood system and endocrine system dysfunction
* noninvasive mechanical ventilation
* active hemoptysis

Min Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xiangyu, MD, Principal Investigator — Shanghai Tebth People's Hospital

REFERENCES:
- [Derived] Wang QX, Zhang XY, Li Q. Effects of a flutter mucus-clearance device on pulmonary function test results in healthy people 85 years and older in China. Respir Care. 2010 Nov;55(11):1449-52. PMID 20979671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recuitment period: April 19th, May 17th location: Redsun geracomium
Groups:
- Intervention Group: all the subjects received portable mucus clearance devices to do pulmonary function rehabilitation.
- Control Group: without any intervention
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 30 | 30
Completed | 27 (3 participants did not complete the period) | 28 (2 participants did not complete the period)
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 30 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 86.81 (2.06) | 87.57 (2.95) | 87.20 (2.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Cases With Fever (Body Temperature Reach 38 Degree Celsius or Higher)
Time Frame: up to 28 days
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 27 | 28
participants | 0 | 2

2. Secondary Outcome: Number of Cases With Antibiotics Therapy
Description: antibiotics therapy is the indicators of pulmonary infection
Time Frame: up to 28 days
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 27 | 28
participants | 1 | 3

3. Primary Outcome: MPEF,Mean Peak Expiratory Flow
Description: indicators of pulmonary function, for example, PEF(unit of measurement:Liter per minute) All subjects sit upright in a chair and instructed to perform the pulmonary function test. Repeat the test until three reproducible acceptable results are obtained. Spirometry was performed at the first day of baseline and the 28th day of our study.
Time Frame: up to 28 days
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 27 | 28
L/min | 117.59 (50.39) | 103.93 (41.53)

4. Primary Outcome: FEV1, Forced Expiratory Volume at First Second
Description: indicators of pulmonary function, for example, FEV1(unit of measurement:Liter)
  All subjects sit upright in a chair and instructed to perform the pulmonary function test. Repeat the test until three reproducible acceptable results are obtained. Spirometry was performed at the first day of baseline and the 28th day of our study.
Time Frame: up to 28 days
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 27 | 28
L | 1.01 (0.37) | 1.02 (0.35)

5. Primary Outcome: FVC, Forced Vital Capacity
Description: indicators of pulmonary function, for example, FVC(unit of measurement:Liter)
  All subjects sit upright in a chair and instructed to perform the pulmonary function test. Repeat the test until three reproducible acceptable results are obtained. Spirometry was performed at the first day of baseline and the 28th day of our study.
Time Frame: up to 28 days
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 27 | 28
L | 2.06 (0.73) | 1.77 (0.63)

6. Primary Outcome: FEV1/FVC%, the Ratio of FEV1 to FVC
Description: indicators of pulmonary function,
  All subjects sit upright in a chair and instructed to perform the pulmonary function test. Repeat the test until three reproducible acceptable results are obtained. Spirometry was performed at the first day of baseline and the 28th day of our study.
Time Frame: up to 28 days
Measure: Mean (Standard Deviation); unit: ratios
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 27 | 28
ratios | 50.67 (16.83) | 59.04 (13.82)

7. Secondary Outcome: Number of Cases With Hospital Visit
Time Frame: up to 28 days
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 27 | 28
participants | 2 | 3

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less